CLINICAL TRIAL: NCT04253119
Title: Retrospective Evaluation of Treatment Durability Among Treatment-naive HIV-infected Individuals Initiated First-line ART in Russia
Brief Title: ART First-line Treatment Durability in Russia
Status: Completed | Type: Observational
Sponsor: MSD Pharmaceuticals LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: VEAP 8370
Record Dates: First submitted 2019-08-02; First posted 2020-02-05 (Actual); Results first posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: HIV-1-infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Antiretroviral/Anti HIV — NNRTI plus two NRTIs or PI boosted by ritonavir with 2 NRTIs per the usual standard of care of the investigator in AIDS clinics of Russia

SUMMARY:
This study is a non-interventional retrospective study. Data from patients who signed informed consent form will be collected through retrospective chart or medical records review. Patients have been receiving treatment and diagnostic procedures according to daily clinical practice conducted by his/her physician. There are no procedures that are required as part of this study.

The study is to be conducted in 6 investigational sites across Russia with up to 200 patients recruited per site.

HIV-infected patients with no experience of therapy at time of initiation of ART with NNRTI plus two NRTIs or PI boosted by ritonavir with 2 NRTIs will be enrolled and followed retrospectively for up to 96 weeks with data collection at the approximate time points of baseline (pre-treatment) and at 48 and 96 weeks after start of treatment.

The following ARV drugs are considered according to the standards of care:

* NNRTIs: efavirenz (EFV), nevirapine (NVP), rilpivirine (RPV), ETR (etravirine)
* PIs: LPV (lopinavir), DRV (darunavir), ATV (atazanavir), FPV (fosamprenavir)

DETAILED DESCRIPTION:
All patients must have initiated ART between February 01 and April 30, 2017. A time window for the retrospective visits at baseline, 48 and 96 weeks is envisaged as approximately ± 8 weeks.

Patients will be retrospectively screened and selected according to inclusion and exclusion criteria prior to enrollment in each investigational site starting the day of its initiation. The study sites will maintain a list of all screened patients. All patients eligible according to the inclusion/exclusion criteria and after signing the informed consent form are to be consequently enrolled for their demographic and clinical data collection through retrospective chart or medical records review. The enrollment will continue until the recruitment goal is reached.

Baseline and follow-up data will be extracted through retrospective chart or medical records review, if available at each investigational site. No additional interventional testsor medical procedures such as additional blood samples, X-ray or other technical investigations will be performed as a part of this study. If any data element is not available, it will be reported as missing.

At baseline, demographic and clinical data on age, gender, employment status, marital status, substance abuse, HIV diagnosis duration, route of infection, AIDS stage, viral load, CD4 count, concomitant medication, comorbidities (noted diagnosis by physician) are to be collected through retrospective chart or medical records review.

At 48 and 96 weeks of retrospective follow-up, the investigators will assess through the medical records whether the patient was still on treatment with initiated ART (NNRTI, PI) and evaluate the estimated time on therapy without change of the NNRTI or PI agent within the class or without change of the NNRTI or PI agent to a different class.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18 years of age) with definite HIV-1 infection based on positive lab test and judgement of treating physician according to standards of care
* Naive to antiretroviral treatment at the time of initiation
* Viral load of >1000 copies/ml at the time of initiation of ART
* Initiated their first-line ART between February 01 and April 30, 2017
* Patients are included, if the third component of their first line ART was either NNRTI or boosted PI plus NRTIs
* Completed follow-up from baseline for at least 96 weeks
* Signed informed consent

Exclusion Criteria:

• HIV-2 infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients enrolled must be treatment naive at the time of initiation of ART with NNRTI plus two NRTIs or PI boosted by ritonavir with 2 NRTIs per the usual standard of care of the investigator in AIDS clinics of Russia.
Sampling Method: Non-Probability Sample
Enrollment: 536 (Actual)
Dates: Start 2019-11-26 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ekaterina Lukyanova, MD, Study Director — MSD Pharmaceuticals LLC
Locations (4):
- Russia (4):
  - Irkutsk Regional AIDS Center, Irkutsk
  - Moscow City AIDS Center of the Moscow Health Department, Moscow
  - Saint-Petersburg AIDS and Infectious Diseases Center, Saint Petersburg
  - Samara Region AIDS Center, Samara

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in investigational sites across Russia with up to 200 patients recruited per site. Each investigational site will be a dedicated HIV clinic or an HIV department in clinic of infectious diseases. It is planned that the first half of the study population (500 patients) will be enrolled during the first 6-9 months and the second half of the study population (500 patients) during the second 6-9 months of the study.
Pre-assignment Details: 536 subjects were enrolled instead of planned 1000 participants due to slow recruitment because of COVID-19 pandemia. This protocol deviation was documented accordingly.
Groups:
- Treatment-naive at the Time of Initiation of ART Per the Usual Standard of Care.: HIV-infected patients with no experience of therapy at time of initiation of ART with NNRTI plus two NRTIs or PI boosted by ritonavir with 2 NRTIs will be enrolled and followed retrospectively for up to 96 weeks with data collection at the approximate time points of baseline (pre-treatment) and at 48 and 96 weeks after start of treatment of the investigator in AIDS clinics of Russia. All patients must have initiated ART between February 01 and June 30, 2017.
Period: Overall Study
Arm/Group | Treatment-naive at the Time of Initiation of ART Per the Usual Standard of Care.
Started | 536
Completed | 536
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment-naive at the Time of Initiation of ART Per the Usual Standard of Care.
Number analyzed (Participants) | 536
Age, Customized [Count of Participants; unit: Participants]
  < 40 years | 338
  40 - 60 years | 187
  > 60 years | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 217
  Male | 319
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Russia | 536

OUTCOME MEASURES:

1. Primary Outcome: 48 Weeks Treatment Durability
Description: Percentage of patients remained on initial therapy without change of the NNRTI or PI agent
Time Frame: 48 weeks
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment-naive at the Time of Initiation of ART Per the Usual Standard of Care.
Number analyzed (Participants) | 536
percentage of participants | 76.0 [72.2 to 79.6]

2. Secondary Outcome: 96 Weeks Treatment Durability
Description: Percentage of patients remained on initial therapy without change of the NNRTI or PI agent
Time Frame: 96 weeks
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment-naive at the Time of Initiation of ART Per the Usual Standard of Care.
Number analyzed (Participants) | 536
percentage of participants | 60.3 [56.0 to 64.4]

3. Secondary Outcome: Time on Therapy at 48 Weeks
Description: Estimated time on therapy without change of the NNRTI or PI agent at 48 weeks among treatment naive HIV-infected individuals initiated ART (NNRTI, PI)
Time Frame: 48 weeks
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Treatment-naive at the Time of Initiation of ART Per the Usual Standard of Care.
Number analyzed (Participants) | 536
weeks | 46.8 (15.1)

4. Secondary Outcome: Time on Therapy at 96 Weeks
Description: Estimated time on therapy without change of the NNRTI or PI agent at 96 weeks among treatment naive HIV-infected individuals initiated ART (NNRTI, PI)
Time Frame: 96 weeks
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Treatment-naive at the Time of Initiation of ART Per the Usual Standard of Care.
Number analyzed (Participants) | 536
weeks | 78.8 (33.8)

ADVERSE EVENTS:
Time Frame: Up to 78 weeks (November 2019 - April 2021)
Arm/Group | Treatment-naive at the Time of Initiation of ART Per the Usual Standard of Care.
All-Cause Mortality (participants affected / at risk) | 0/536
Serious Adverse Events (participants affected / at risk) | 0/536
Other Adverse Events (participants affected / at risk) | 0/536

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-02): https://cdn.clinicaltrials.gov/large-docs/19/NCT04253119/Prot_SAP_000.pdf